CLINICAL TRIAL: NCT05322837
Title: Deep Phenotyping of Upper Limb Sensori-motor Recovery in Asian Stroke Survivors: Concept, Development and Implementation of a Rehabilomics-driven Technology-assisted Data Platform
Brief Title: Tracking of Upper Limb Sensory and Motor Recovery in Asian Stroke Survivors
Status: Recruiting | Type: Observational
Sponsor: Tan Tock Seng Hospital (Other)
Collaborators: Rehabilitation Research Institute of Singapore (RRIS) (Unknown); Singapore-ETH Centre (SEC) (Unknown)
Responsible Party: Sponsor
Other Study IDs: DSRB 2021/00919
Record Dates: First submitted 2022-04-01; First posted 2022-04-12 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Intervention
  Interventions: Other: Clinical and technological-aided assessments and questionnaires

INTERVENTIONS:
Other: Clinical and technological-aided assessments and questionnaires — Assessments and questionnaires related to upper limb function and quality of life will be used

SUMMARY:
As Singapore's population is aging rapidly, the incidence rate of stroke has been increasing in the past years. Rehabilitation is essential for the resumption of daily activities, and with the appropriate care, it is possible for stroke-survivors to regain most of their functions.

Hence, this study aims to better understand upper limb recovery covering different stages post-stroke in a representative cohort of Asian adults

DETAILED DESCRIPTION:
Stroke is a leading contributor to disability in Singapore, partially driven by a reduced ability to use the upper limb in their daily lives. Reduced upper limb use commonly results from a variety of impairments such as motor, sensory and cognitive impairments.

The aim of this longitudinal and observational study is to gather a rich multi-modal database on the time-course of upper limb recovery in a representative cohort after stroke and characterise the relationship between upper limb recovery, common post-stroke impairments and quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. Stroke confirmed by neurologists, neurosurgeons and brain imaging (CT, CT angiogram, MRI, MR angiogram)
2. First ever confirmed stroke
3. Asian ethnicity
4. Age 21-90 years
5. Montreal Cognitive Assessment (MOCA) scores 21/30 and above
6. Admission to rehabilitation ward is within 8 weeks of stroke onset

Exclusion Criteria:

1. Recurrent stroke or transient ischaemic attack (TIA)
2. Upper limb impairment not related to stroke: e.g., subarachnoid haemorrhage, traumatic brain injury or brain tumours
3. Bilateral upper limb impairment.
4. Uncontrolled medical conditions such as hypertension, hypotension, diabetes mellitus, unstable angina, cardiac failure or sepsis will be excluded.
5. Active fractures or arthritis of upper limb joints/bones
6. Visual Analogue Scale (VAS) pain > 5/10
7. MOCA < 21/30
8. Severe behavioural disturbance or agitation or epilepsy or untreated depression
9. Life expectancy < 6 months
10. End organ failures on replacements (renal dialysis or renal replacement therapies)
11. Minimally responsive or unresponsive awareness (vegetative) states
12. Pregnancy or lactation states
13. Admission to rehab ward later than 8 weeks post-stroke
14. (For TMS assessments only) History of epilepsy or seizures, or cranial surgeries, or have metal implants in body or head, or have implanted electronics, or have metallic valve, or skull fracture or brain injury, or head or brain surgeries.

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to inpatient rehabilitation unit
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2023-04-26 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Fugl-Meyer Assessment (FMA) | Inpatient: week 1 of admission
  The FMA-UE is a stroke-specific, performance-based impairment index. It is designed to assess motor functioning, balance, in patients with post-stroke hemiplegia.

CONTACTS AND LOCATIONS:
Overall Officials: Dr Karen Chua, MBBS, Principal Investigator — Tan Tock Seng Hospital
Locations (1):
- Tan Tock Seng Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cheng HJ, Chin LF, Kanzler CM, Lehner R, Kuah CWK, Kager S, Josse E, Samkharadze T, Sidarta A, Gonzalez PC, Lie E, Zbytniewska-Megret M, Wee SK, Liang P, Gassert R, Chua K, Lambercy O, Wenderoth N. Upper limb sensorimotor recovery in Asian stroke survivors: a study protocol for the development and implementation of a Technology-Assisted dIgitaL biOmaRker (TAILOR) platform. Front Neurol. 2023 Nov 30;14:1246888. doi: 10.3389/fneur.2023.1246888. eCollection 2023. PMID 38107648